CLINICAL TRIAL: NCT02390453
Title: Cognitive and Aerobic Resilience for the Brain
Acronym: CARB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Frederick Unverzagt, Professor, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: R01AG045157 (NIH); 1R01AG045157-01A1 (NIH)
Record Dates: First submitted 2015-03-05; First posted 2015-03-17 (Estimated); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Mild Cognitive Impairment
Keywords: mild cognitive impairment; randomized controlled trial; cognitive training; exercise training; cognition; physical performance; disability; mood
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Restraint, Physical

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Combined Cognitive and Physical (Experimental): This consists of 45 minutes of Cognitive arm + 45 minutes of Physical arm (90 minutes total), 3 days a week for 12 weeks (36 sessions).
  Interventions: Behavioral: Combined Cognitive and Physical
- Cognitive (Active Comparator): This consists of 45 minutes of cognitive modules from Posit Science, 3 days a week for 12 weeks (36 sessions).
  Interventions: Behavioral: Cognitive
- Physical (Active Comparator): This consists of 45 minutes of multi-modal physical exercise, 3 days a week for 12 weeks (36 sessions).
  Interventions: Behavioral: Physical
- Active Control (Active Comparator): This consists of 45 minutes of group discussion of health and successful aging, 2 days a week for 12 weeks (24 sessions).
  Interventions: Behavioral: Active Control

INTERVENTIONS:
Behavioral: Combined Cognitive and Physical — Combined modules provide Cognitive training from Posit Science designed to improve information processing speed, learning, memory, and attention, and Physical training focused on seated aerobic and progressive resistance exercises designed to improve aerobic capacity, muscular strength, and endurance consistent with current exercise recommendations for older adults.
  Arms: Combined Cognitive and Physical
Behavioral: Cognitive — Cognitive modules from Posit Science are designed to improve information processing speed, learning, memory, and attention.
  Arms: Cognitive
Behavioral: Physical — Physical modules are focused on seated aerobic and progressive resistance training designed to improve aerobic capacity, muscular strength, and endurance consistent with current exercise recommendations for older adults.
  Arms: Physical
Behavioral: Active Control — Control modules provide social contact for group discussion of health and successful aging.
  Arms: Active Control

SUMMARY:
This is a randomized controlled trial (RCT) of the effectiveness of cognitive and exercise training versus control condition on cognitive function in older adults with mild cognitive impairment (MCI).

DETAILED DESCRIPTION:
Exercise and cognitive training hold promise for delaying progression of MCI. Exercise improves cognitive ability, brain function, and brain structure in older adults. Cognitive training has been shown to durably improve mental abilities and functional status in older adults. In addition, persons with MCI respond to some forms of cognitive training just as robustly as healthy older adults.

This pilot study is a 4 group design with a home-based multi-modal physical exercise intervention, cognitive training, combined cognitive and physical training, and a social contact control enrolling older adults with MCI.

This pilot study is designed to be consistent with current recommended approaches to establishing trial feasibility. If the aims are achieved, it will provide a conceptual and practical rationale to support a large, multi-site, randomized clinical trial to test the efficacy of combined physical and cognitive training in delaying time to a clinical diagnosis of dementia.

ELIGIBILITY:
Inclusion Criteria:

* subjective memory complaint
* minimal impairment in daily function per Functional Activity Questionnaire (FAQ)
* sedentary
* English speaking
* access to telephone

Exclusion Criteria:

* dementia or Alzheimer disease
* stroke, past 12 months
* myocardial infarction, past 12 months
* angina
* Parkinson disease
* multiple sclerosis
* epilepsy
* AIDS
* brain tumor, infection, or surgery
* brain injury with > 30 minute LOC
* schizophrenia
* bipolar disorder
* cancer with short life expectancy
* current chemotherapy or radiation therapy
* depression
* alcohol consumption ≥ 8 drinks per week for women, or ≥15 drinks per week for men
* prescription of Aricept or Namenda, past or present
* self-reported difficulty reading a newspaper (low visual acuity)
* low hearing or communicative ability (examiner-rated) that would interfere with interventions and outcome assessments
* prior involvement in similar cognitive training studies, programs, or online training
* prior use of online brain training or brain fitness programs
* unable to pass the Exercise Assessment and Screening for You (EASY)
* living in nursing home
* scheduling conflicts with intervention schedule
* unwilling to use a computer or be on video conferencing
* Baseline blood pressure of Systolic > 180
* Baseline blood pressure of Diastolic > 100
* Baseline pulse of < 40 or > 100
* unable to provide informed consent

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 201 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2019-10-25 (Actual); Study Completion 2019-10-25 (Actual)

PRIMARY OUTCOMES:
Cognitive function composite score as measured by individually-administered tests of psychomotor speed, complex sequencing, and list learning. | End of treatment at 12-weeks.
  The cognitive composite is derived from: WAIS-IV Symbol Search, Trail Making Test Part B, and Rey Auditory Verbal Learning Test.
Average participant self-ratings of intervention acceptability. | From date of randomization until the date of the final training session or the end of the 12-week intervention, whichever came first.
  Average of individual Likert self-ratings of the interventions (where 1 = very unenjoyable, 2 = not enjoyable, 3 = neutral, 4 = enjoyable, and 5 = very enjoyable) for each session of the 12-week intervention.
Participant adherence to treatment. | From date of randomization until the date of the final training session or the end of the 12-week intervention, whichever came first.
  Number of training sessions attended divided by the the total number of sessions available.
Participant adherence to outcome assessment. | End of treatment at 12-weeks.
  Number of participants completing the post-training outcome assessment divided by the total number randomized.
Number of participants with study-related adverse events (AE) by treatment arm. | From enrollment through end of treatment at 12-weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Frederick W Unverzagt, PhD, Principal Investigator — Indiana University
Locations (1):
- Indiana University, Indianapolis, Indiana, United States